CLINICAL TRIAL: NCT04056910
Title: Phase II Study of IDH1 Inhibitor Ivosidenib and Nivolumab in IDH1 Mutant Gliomas and Advanced Solid Tumors
Brief Title: Ivosidenib (AG-120) With Nivolumab in IDH1 Mutant Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jason J. Luke, MD (Other)
Collaborators: Agios Pharmaceuticals, Inc. (Industry); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor-Investigator, Jason J. Luke, MD, Associate Professor of Medicine, University of Pittsburgh Medical Center
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCC 19-096
Record Dates: First submitted 2019-08-12; First posted 2019-08-14 (Actual); Results first posted 2025-02-06 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Advanced Solid Tumor; IDH1 Mutation; Glioma
MeSH Terms: conditions — Glioma | interventions — ivosidenib; Nivolumab

STUDY DESIGN:
Intervention Model Description: Concurrent dosing of ivosidenib and nivolumab.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Concurrent dosing of ivosidenib and nivolumab (Experimental): Ivosidenib will be administered concurrently with nivolumab on a Q28 day schedule.
  Interventions: Drug: ivosidenib and nivolumab

INTERVENTIONS:
Drug: ivosidenib and nivolumab — Ivosidenib will be administered orally at a dose of 500 mg (provided as 250 mg strength tablets) daily. The dose may be reduced to 250 mg for patients experiencing more than one event of Grade 2 nausea or vomiting (related or unrelated), or Grade 3 or Grade 4 adverse events. Nivolumab will be administered at 480 mg IV every 28 days.

SUMMARY:
In this study, response to treatment and (progression free and overall) survival will be described and safety events of ivosidenib in combination with nivolumab will be summarized in patients with advanced solid tumors (nonresectable or metastatic) or enhancing gliomas.

DETAILED DESCRIPTION:
This study will describe the safety, response rate, progression free and overall survival, and summarize safety events of ivosidenib in combination with nivolumab in participants with advanced solid tumors (nonresectable or metastatic) or enhancing gliomas. Participants are required to have a histologically consistent diagnosis of IDH1 gene mutated tumor that is not eligible for curative therapy. Enrolled subjects will receive orally administered ivosidenib dosed daily on 28-day cycles and nivolumab will be infused every 28 days. Participants will be assessed at every visit for adverse events starting from the first dose of study treatment. Assessment (CT or MRI) for evaluation of disease response will be conducted every 8 weeks (±7 days) from the first day of treatment cycle 1 and/or at any time when progression of disease is suspected. A Post-Treatment Follow-Up Visit for safety will occur 28 (+/- 5) days after the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Be ≥18 years of age.
* Have a histopathological diagnosis (fresh or banked tumor biopsy sample, preferably collected within the last 3 years) of an advanced solid tumor for which curative treatment is not available and have undergone appropriate standard of care treatment options (in the opinion of the treating investigator).
* Have a documented IDH1 gene-mutated disease (from a fresh tumor biopsy or the most recent banked tumor tissue available) based on CLIA certified sequencing (R132C/L/G/H/S mutation variants tested).

  * For glioma, must have both 1) contrast enhancing disease and 2) WHO 2016 grade II
* Have an ECOG PS score of 0 or 1 (Appendix 11.1)
* Have at least one evaluable and measurable lesion as defined by RECIST v1.1 (solid tumors) or Response Assessment in Neuro-Oncology (RANO) Criteria (glioma).
* Have recovered from toxicities associated with prior anticancer therapy to baseline or ≤ grade 1 unless stabilized under medical management per investigator.
* Have adequate bone marrow function as evidenced by:

  * Absolute neutrophil count ≥ 1,500/mm3 or 1.5 × 109/L
  * Hemoglobin ≥ 8 g/dL
  * Platelets ≥ 100,000/mm3 or 100 × 109/L
* Have adequate hepatic function as evidenced by:

  * Serum total bilirubin ≤ 2 × upper limit of normal (ULN), unless considered due to Gilbert's disease
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 5 × ULN in the presence of liver metastases (or primary hepatic tumor) OR ≤ 2× ULN within glioma patients
* Have adequate renal function as evidenced by:

  • Serum creatinine < 1.5 × ULN OR Creatinine clearance ≥ 50 mL/min based on the Cockroft-Gault glomerular filtration rate (GFR) estimation: (140 - Age) x (weight in kg) x (0.85 if female)/72 x serum creatinine
* Be able to understand and willing to sign the informed consent form (or have legal representation) and to comply with scheduled visits, treatment plans, procedures, and laboratory tests, including serial peripheral blood sampling, biopsies, and urine sampling, during the study. A legally authorized representative may consent on behalf of a participant who is otherwise unable to provide informed consent if acceptable to and approved by the IRB/Independent Ethics Committee (IEC).
* Female participants with reproductive potential must have negative serum pregnancy testing within 72 h prior to the initial administration of study drug, then every 4 weeks±1 week, or a negative confirmation from an obstetrician in case of equivocal serum pregnancy results. Females of reproductive potential are defined as sexually mature women who have not undergone a hysterectomy, bilateral oophorectomy, or tubal occlusion or who have not been naturally postmenopausal (ie, who have not menstruated) for at least 24 consecutive months (ie, have not had menses at any time in the preceding 24 consecutive months). Men with partners who are women with reproductive potential must agree that they or their partners will use two effective forms of contraception (including at least one barrier form) when engaging in reproductive sexual activity.
* Women of child-bearing potential (WOCBP) receiving nivolumab will be instructed to adhere to contraception for a period of 5 months after the last dose of nivolumab. Men receiving nivolumab and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 7 months after the last dose of nivolumab.
* Effective forms of contraception are defined as hormonal oral contraceptives, injectables, patches, intrauterine devices, intrauterine hormone-releasing systems, bilateral tubal ligation, condoms with spermicide, or male partner sterilization.

Exclusion Criteria:

* Received a prior IDH inhibitor.
* Received systemic anticancer therapy or an investigational agent < 2 weeks prior to Day 1). In addition, the first dose of study treatment should not occur before a period ≥ 5 half-lives (t1/2)of the investigational agent has elapsed.
* For solid tumor patients: received radiotherapy to metastatic sites of disease < 2 weeks prior to Day 1 and for glioma patients have received radiation within 3 months prior.
* For solid tumor patients, have underwent hepatic radiation, chemoembolization, and radiofrequency ablation < 4 weeks prior to Day 1.
* Participants must not have a diagnosis of immunodeficiency or is receiving systemic steroid therapy at a dose of > 10 mg prednisone daily or equivalent at time of first dose of study treatment.
* Participants must not have active autoimmune disease that has required systemic treatment in the past 2 years (ie, with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroids replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Participants must not have a known history of non-infectious pneumonitis that required steroids for treatment.
* Participants must not have evidence of interstitial lung disease.
* For solid tumor patients, have known symptomatic brain metastases requiring steroids. Participants with previously diagnosed brain metastases are eligible if they have completed their treatment and have recovered from the acute effects of radiation therapy or surgery prior to study entry, have discontinued corticosteroid treatment for these metastases for at least 1 week and have radiographically stable disease for at least 1 month prior to study entry.
* Have a history of another primary cancer that is active requiring treatment, progressing or for which the treating investigator believes will make disease assessment unreliable.
* Have evidence of intracranial or intra-tumoral hemorrhage either by MRI or computed tomographic (CT) scan. Participants with resolving post-surgical changes, punctate hemorrhage, or hemosiderin are eligible.
* Underwent major surgery within 4 weeks of Day 1 or have not recovered from post-surgery toxicities.
* Are pregnant or breastfeeding.
* Are taking known strong CYP3A4 inducers or sensitive CYP3A4 substrate medications with a narrow therapeutic window (Appendix 0), unless they can be transferred to other medications within ≥5 t1/2 prior to dosing.
* Are taking P-glycoprotein (P-gp) transporter-sensitive substrate medications with a narrow therapeutic window (Appendix 0), unless they can be transferred to other medications within ≥ 5 t1/2 prior to administration of study treatment.
* Have an active infection requiring systemic anti-infective therapy or with an unexplained fever > 38.5°C within 7 days of Day 1 (at the discretion of the treating investigator) participants with tumor fever may be enrolled).
* Have any known hypersensitivity to any of the components of ivosidenib or nivolumab.
* Have significant active cardiac disease within 6 months prior to the start of study treatment, including New York Heart Association (NYHA) Class III or IV congestive heart failure (Appendix 0); myocardial infarction; unstable angina; and/or stroke.
* Have a heart-rate corrected QT interval (using Fridericia's formula) (QTcF) (Appendix 0) ≥ 480 ms or other factors that increase the risk of QT prolongation or arrhythmic events (eg, heart failure, hypokalemia, family history of long QT interval syndrome). Bundle branch block and prolonged QTcF interval are permitted with approval of the Medical Monitor.
* Are taking medications that are known to prolong the QT interval (Appendix 0), unless they can be transferred to other medications within ≥ 5 t1/2 prior to dosing or unless the medications can be properly monitored during the study. (If equivalent medication is not available, QTcF should be closely monitored.)
* Have known active hepatitis B (HBV) or hepatitis C (HCV) infections, known positive human immunodeficiency virus (HIV) antibody results, or acquired immunodeficiency syndrome (AIDS) related illness. Participants with a sustained viral response to HCV treatment or immunity to prior HBV infection will be permitted. Participants with chronic HBV that is adequately suppressed per institutional practice will be permitted.
* Have any other acute or chronic medical or psychiatric condition, including recent (within 12 months of Day 1) or active suicidal ideation or behavior, or a laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the treating investigator, would make the participant inappropriate for entry into this study.
* Have known active inflammatory gastrointestinal disease, chronic diarrhea, previous gastric resection or lap band dysphagia, short-gut syndrome, gastroparesis, or other conditions that limit the ingestion or gastrointestinal absorption of drugs administered orally. Gastroesophageal reflux disease under medical treatment is allowed (assuming no drug interaction potential).
* Have been committed to an institution by an order issued either by the judicial or administrative authorities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-09-20 (Actual); Primary Completion 2023-11-13 (Actual); Study Completion 2023-11-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason J Luke, MD, PhD, Principal Investigator — UPMC Hillman Cancer Center
Locations (1):
- UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nguyen MK, Jelinek M, Singh A, Isett B, Myers ES, Mullett SJ, Eisele Y, Beumer JH, Parise RA, Urban J, Rose A, Sellitto L, Singh K, Doerfler R, Dadey RE, Kim C, Rhee JC, Davar D, Villaruz LC, Burgess M, Drappatz J, Mantica M, Goodman AE, Wang H, Singhi AD, Luke JJ, Zandberg DP, Bao R. Clinical and translational study of ivosidenib plus nivolumab in advanced solid tumors harboring IDH1 mutations. Oncologist. 2025 Nov 11;30(11):oyaf362. doi: 10.1093/oncolo/oyaf362. PMID 41138165
- [Derived] Nguyen MK, Jelinek M, Singh A, Isett B, Myers ES, Mullett SJ, Eisele Y, Beumer J, Parise R, Urban J, Rose A, Sellitto L, Singh K, Doerfler R, Dadey RE, Kim C, Rhee JC, Davar D, Villaruz LC, Burgess M, Drappatz J, Mantica M, Goodman AE, Wang H, Singhi AD, Luke JJ, Zandberg DP, Bao R. Clinical and translational study of ivosidenib plus nivolumab in advanced solid tumors harboring IDH1 mutations. medRxiv [Preprint]. 2025 Jul 21:2025.07.19.25331848. doi: 10.1101/2025.07.19.25331848. PMID 40778139

RESULTS

PARTICIPANT FLOW:
Groups:
- Concurrent Dosing of Ivosidenib and Nivolumab: Ivosidenib will be administered concurrently with nivolumab on a Q28 day schedule.
  ivosidenib and nivolumab: Ivosidenib will be administered orally at a dose of 500 mg (provided as 250 mg strength tablets) daily. The dose may be reduced to 250 mg for patients experiencing more than one event of Grade 2 nausea or vomiting (related or unrelated), or Grade 3 or Grade 4 adverse events.
  Nivolumab will be administered at 480 mg IV every 28 days.
Period: Overall Study
Arm/Group | Concurrent Dosing of Ivosidenib and Nivolumab
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All study-eligible participants
Arm/Group | Concurrent Dosing of Ivosidenib and Nivolumab
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.13 (12.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
ECOG Performance Score [Count of Participants; unit: Participants] — 0 = Fully active; no restrictions
  1. = Restricted in strenuous activity; able to do light/sedentary work
  2. = Capable of selfcare; physically active 50% of awake hours
  3. = Limited selfcare ability; confined to bed or chair during 50% of awake hours
  4. = Fully disabled; Unable to do selfcare; totally confined to bed/chair
  Participants
    ECOG Performance Score = 0 | 6
    ECOG Performance Score = 1 | 9
Disease Site [Count of Participants; unit: Participants] — Anatomical site of primary disease
  Participants
    BILE DUCT - INTRAHEPATIC | 1
    BILIARY TRACT - NOS | 1
    BONES - NOS | 1
    BONES - RIB STER CLAV & ASS JTS | 1
    BRAIN - FRONTAL LOBE | 1
    BRAIN - NOS | 5
    BRAIN - PARIETAL LOBE | 1
    COLON - DESCENDING | 1
    GALLBLADDER | 2
    SKIN - UPPER LIMB AND SHOULDER | 1
Histology [Count of Participants; unit: Participants] — Histology type of primary disease site
  Participants
    ADENOCARCINOMA, N/A | 1
    ASTROCYTOMA, ANAPLASTIC | 1
    ASTROCYTOMA, NOS | 2
    CARCINOMA, METASTATIC, NOS | 1
    CHOLANGIOCARCINOMA | 2
    CHONDROSARCOMA, NOS | 1
    CHONDROSARCOMA, NOS, MAL, MET | 1
    GLIOBLASTOMA, NOS | 1
    NEOPLASM, MALIGNANT | 2
    OLIGODENDROGLIOMA, ANAPLASTIC | 2
    OLIGODENDROGLIOMA, NOS | 1

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Response
Description: Number of patients with Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (target or non-target) with reduction in short axis to <10 mm, Partial Response (PR): ≥30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters or Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters per RECIST v1.1 Criteria, or, per RANO Criteria: Complete Response (CR): Observed in consecutive assessments ≥4 weeks apart per RANO. Partial Response (PR): Observed in consecutive assessments ≥4 weeks apart per RANO.
Time Frame: At 8 weeks after first treatment; up to 14 months for cohort
Population: Patients who received treatment and were evaluated for radiologic response.
Measure: Count of Participants; unit: Participants
Arm/Group | Concurrent Dosing of Ivosidenib and Nivolumab
Number analyzed (Participants) | 7
Participants
  Partial Response (PR) | 1
  Stable Disease (SD) | 6

2. Primary Outcome: Six Month Progression-Free Survival (PFS6)
Description: Percentage of participants surviving without objective tumor progression at six months after the initiation of treatment.
  Per RECIST v1.1 Criteria: Progressive Disease (PD): ≥20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). The sum must also demonstrate an absolute increase of ≥5 mm. The appearance ≥1 new lesion(s) is considered progression.
  Per RANO Criteria: Progressive Disease: No CR, PR, SD prior to PD. Progression: 25% or more increase in enhancing lesions despite stable or increasing steroid dose, increase (significant) in non-enhancing FLAIR/T2W lesions, not attributable to other non-tumor causes, any new lesions; clinical deterioration (not attributable to other non-tumor causes and not due to steroid decrease)
Time Frame: At 6 months
Population: Patients who received treatment and were evaluated for radiologic response who did not experience disease progression at the designated time frame.
Measure: Number; unit: percentage of participants
Arm/Group | Concurrent Dosing of Ivosidenib and Nivolumab
Number analyzed (Participants) | 15
percentage of participants | 20

3. Secondary Outcome: Occurrence of Dose Limiting Toxicity (DLT)
Description: The occurrence (number) of dose limiting toxicity (DLT) in patients receiving ivosidenib plus nivolumab. DLT describes side effects of the treatment that are serious enough to prevent an increase in dose or level of that treatment. CTCAE v5 was used to assess Adverse Events and Serious Adverse Events.
Time Frame: Up to 24 months
Population: Treated patients assessed for Dose Limiting Toxicities.
Measure: Count of Participants; unit: Participants
Arm/Group | Concurrent Dosing of Ivosidenib and Nivolumab
Number analyzed (Participants) | 15
Participants | 0

4. Secondary Outcome: Adverse Events Related to Treatment
Description: Number of patients who experienced Adverse Events or Serious Adverse Events per NCI Common Terminology Criteria for Adverse Events (CTCAE v5.0), that were related to their receiving the treatment combination of ivosidenib and nivolumab.
Time Frame: Up to 24 months
Population: Patients who experienced a treated-related adverse event.
Measure: Count of Participants; unit: Participants
Arm/Group | Concurrent Dosing of Ivosidenib and Nivolumab
Number analyzed (Participants) | 13
Participants
  Anemia | 2
  Eosinophilia | 1
  QTC prolongation | 2
  Thyroid Stimulating Hormone Increased | 3
  Hypothyroidism | 4
  Diarrhea | 4
  Nausea | 1
  Vomiting | 2
  Fatigue | 1
  Flu like symptoms | 1
  Weight loss | 1
  Infusion related reaction | 2
  Alanine aminotransferase increased | 1
  Aspartate aminotransferase increased | 1
  Blood bilirubin increased | 1
  Lymphocyte count decreased | 2
  Neutrophil count decreased | 2
  Anorexia | 1
  Arthralgia | 1
  Gait disturbance | 1
  Hip pain | 1
  Muscle cramps- intermittent | 1
  Pruritus | 3
  Rash maculo-papular | 9
  Rash | 1
  Hyperthyroidism | 1

5. Secondary Outcome: Progression Free Survival (PFS)
Description: The time from first dose of either drug until disease progression or death from any cause, whichever occurs first.
  RECIST v1.1 Criteria: Progressive Disease (PD): ≥20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). The sum must also demonstrate an absolute increase of ≥5 mm. The appearance ≥1 new lesion(s) is considered progression.
  RANO Criteria: Progressive Disease: No CR, PR, SD prior to PD. Progression: 25% or more increase in enhancing lesions despite stable or increasing steroid dose, increase (significant) in non-enhancing FLAIR/T2W lesions, not attributable to other non-tumor causes, any new lesions; clinical deterioration (not attributable to other non-tumor causes and not due to steroid decrease)
Time Frame: Up to 25 months
Population: Patients who received treatment and were evaluated for radiologic response and who did not experience disease progression during the designated time frame.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Concurrent Dosing of Ivosidenib and Nivolumab
Number analyzed (Participants) | 15
months | 1.94 [1.61 to 3.68]

ADVERSE EVENTS:
Time Frame: All-Cause Mortality - up to 25 months Serious Adverse Events and Adverse Events - up to 24 months (population)
Arm/Group | Concurrent Dosing of Ivosidenib and Nivolumab
All-Cause Mortality (participants affected / at risk) | 1/15
Serious Adverse Events (participants affected / at risk) | 4/15
Other Adverse Events (participants affected / at risk) | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Concurrent Dosing of Ivosidenib and Nivolumab (N=15)
Atrial fibrillation (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Hyperthyroidism (Endocrine disorders) | 1
Flashing lights (Eye disorders) | 1
Catheter related infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Concurrent Dosing of Ivosidenib and Nivolumab (N=15)
Anemia (Blood and lymphatic system disorders) | 7
Eosinophilia (Blood and lymphatic system disorders) | 1
Coronary artery disease (Cardiac disorders) | 1
QTC prolongation (Cardiac disorders) | 4
Sinus tachycardia (Cardiac disorders) | 3
Thyroid Stimulating Hormone Increased (Endocrine disorders) | 5
Hyperthyroidism (Endocrine disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Double Vision - Intermittent (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Bloating (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 8
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 2
Fatigue (General disorders) | 7
Fever (General disorders) | 2
Flu like symptoms (General disorders) | 1
Gait disturbance (General disorders) | 1
Ascites (General disorders) | 1
Weight loss (General disorders) | 2
Infusion related reaction (General disorders) | 1
Localized edema (General disorders) | 1
Pain (General disorders) | 1
Sinusitis (Infections and infestations) | 1
Wound infection (Infections and infestations) | 1
Activated partial thromboplastin time prolonged (Investigations) | 1
Alanine aminotransferase increased (Investigations) | 3
Alkaline phosphatase increased (Investigations) | 4
Aspartate aminotransferase increased (Investigations) | 3
Blood bilirubin increased (Investigations) | 3
Creatinine increased (Investigations) | 1
Blood Lactate Dehydrogenase Increased (Investigations) | 8
Blood Lactate Dehydrogenase Increased (intermittent) (Investigations) | 1
Lymphocyte count decreased (Investigations) | 7
Neutrophil count decreased (Investigations) | 6
Platelet count decreased (Investigations) | 2
Weight gain (Investigations) | 2
Weight loss (Investigations) | 2
White blood cell decreased (Investigations) | 4
Anorexia (Metabolism and nutrition disorders) | 2
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 4
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hyperuricemia (Metabolism and nutrition disorders) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 2
Hypocalcemia (Metabolism and nutrition disorders) | 2
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 3
Hyponatremia (Metabolism and nutrition disorders) | 6
Hypophosphatemia (Metabolism and nutrition disorders) | 5
Hyperphosphatemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2
Gait disturbance (Musculoskeletal and connective tissue disorders) | 1
Hip pain (Musculoskeletal and connective tissue disorders) | 1
Left Calf Pain (Musculoskeletal and connective tissue disorders) | 1
Muscle cramps- intermittent (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Memory impairment (Nervous system disorders) | 2
Dizziness - Intermittent (Nervous system disorders) | 1
Epileptic Aphasia (Nervous system disorders) | 1
impaired concentration (Nervous system disorders) | 1
impaired short term memory (Nervous system disorders) | 1
Nystagmus (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 1
Panic Attacks (Intermittent) (Psychiatric disorders) | 1
Chronic kidney disease (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 2
Nocturnal enuresis (Renal and urinary disorders) | 1
UTI (Renal and urinary disorders) | 1
Urine discoloration (Renal and urinary disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 9
Excessive Dryness - Feet (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Rash - Right Hand (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-01): https://cdn.clinicaltrials.gov/large-docs/10/NCT04056910/Prot_SAP_000.pdf